CLINICAL TRIAL: NCT01264549
Title: Stroke Adverse Outcome is Associated With Nosocomial Infections: PCTus- Guided Antibacterial Therapy in Severe Ischemic Stroke Patients
Brief Title: Stroke Adverse Outcome is Associated With Nosocomial Infections: PCTus- Guided Antibacterial Therapy in Severe Ischemic Stroke Patients (STRAWINSKI)
Acronym: STRAWINSKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Brahms AG (Industry); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. Andreas Meisel, Charité University, Berlin, Germany (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC), Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STRAWINSKI
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; stroke-associated infections; biomarkers; PCT; immune and infection parameters
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCT guided arm (Experimental)
  Interventions: Device: Procalcitonin assay - B.R.A.H.M.S PCT ultrasensitive Kryptor
- Control (No Intervention): Standard treatment

INTERVENTIONS:
Device: Procalcitonin assay - B.R.A.H.M.S PCT ultrasensitive Kryptor — The physician will be given access to a PCT value for Day 1 - 7. Depending on the PCT concentrations, the protocol recommends or discourages from the use of antibiotics
  Other Names: Procalcitonin
  Arms: PCT guided arm

SUMMARY:
Development of stroke associated pneumonia (SAP) has a detrimental effect on stroke outcome. Biomarker-guided antibiotic treatment of patients at high risk for pneumonia may help to improve stroke outcome. Therefore, the investigators will evaluate whether intensified infection monitoring via Procalcitonin guiding an early standardized antibiotic treatment improves functional outcome after stroke compared with standard therapy based on current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* stroke onset within the last 40 hours before randomisation
* clinical diagnosis of a severe (NIHSS > 9), non-lacunar stroke in the middle cerebral artery territory
* consent given by the patient or by his/her legitimate representative where patients are incapable of giving consent themselves

Exclusion Criteria:

* CT evidence of an intracerebral haemorrhage or a lacunar infarct as the probable cause of the current illness
* Antibiotic use within the last 10 days
* Suspected life expectancy of < 3 months
* Participation in other interventional trials (on pharmaceuticals or medical devices)
* Pregnancy, lactation
* Pre-stroke mRS score ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS 0-6) score 0-4 adjusted for baseline modified Rankin score | 3 months after onset of symptoms (stroke)
  To assess the proportion of patients with a modified Rankin scale (mRS 0-6) score 0-4 at day 90 adjusted for baseline modified Rankin score.

SECONDARY OUTCOMES:
Proportion of patients receiving any antibiotic therapy | 3 months after onset of symptoms (stroke)
  To assess the proportion of patients receiving any antibiotic therapy for any duration within 90 days.
Modified Rankin scale adjusted for baseline modified Rankin score | 3 months after onset of symptoms (stroke)
  To assess the Modified Rankin scale at day 90 adjusted for baseline modified Rankin score.
Barthel Index adjusted for baseline Barthel Index | 3 months after onset of symptoms (stroke)
  To assess the Barthel Index (BI 0-100) at day 90 adjusted for baseline Barthel Index.
Modified Rankin scale (mRS) score 0-4 adjusted for baseline modified Rankin score | 6 months after onset of symptoms (stroke)
  To assess the proportion of patients with a modified Rankin scale (mRS) score 0-4 at day 180 adjusted for baseline modified Rankin score.
Modified Rankin scale adjusted for baseline modified Rankin score | 6 months after onset of symptoms (stroke)
  To assess the modified Rankin scale at day 180 adjusted for baseline modified Rankin score.
Barthel Index adjusted for baseline Barthel Index | 6 months after onset of symptoms (stroke)
  To assess the Barthel Index at day 180 adjusted for baseline Barthel Index.
Days alive and out of hospital | 3 months after onset of symptoms (stroke)
  To assess the days alive and out of hospital at day 90.
Time to first event of death, re-hospitalization or recurrent stroke | within 6 months after onset of symptoms (stroke)
  To assess the time to first event of death, re-hospitalization or recurrent stroke.
Proportion of events of post stroke infections | within 7 days after onset of symptoms (stroke)
  To assess the proportion of events of post stroke infections to day 7.
Proportion of events of post stroke infection or death | within 7 days after onset of symptoms (stroke)
  To assess the proportion of events of post stroke infection or death to day 7.
Medium number of days with fever (≥ 37,5°C) per patient | within 7 days after onset of symptoms (stroke)
  To assess the medium number of days with fever (≥ 37,5°C) per patient to day 7.
Stroke volume analysis | 6 months after onset of symptoms (stroke)
  To investigate the effect of an early PCT-guided antiinfective therapy on stroke volume.
Length of hospital stay | on discharge
  To assess the length of hospital stay after acute stroke.
Hospital discharge disposition | on discharge
  To assess the disposition on hospital discharge.
shift analysis of the mRS

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charité University Berlin (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC); Stefan Anker, MD PhD, Principal Investigator — Charité University Berlin (Dept of Cardiology)
Locations (6):
- Germany (5):
  - Charite University (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC), Berlin
  - Unfallkrankenhaus Berlin Neurologie, Berlin
  - Vivantes Auguste Viktoria Klinikum Neurologie, Berlin
  - Vivantes Neukölln Neurologie, Berlin
  - Klinikum Frankfurt (Oder) Neurologie, Frankfurt (Oder)
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Ulm L, Hoffmann S, Nabavi D, Hermans M, Mackert BM, Hamilton F, Schmehl I, Jungehuelsing GJ, Montaner J, Bustamante A, Katan M, Hartmann A, Ebmeyer S, Dinter C, Wiemer JC, Hertel S, Meisel C, Anker SD, Meisel A. The Randomized Controlled STRAWINSKI Trial: Procalcitonin-Guided Antibiotic Therapy after Stroke. Front Neurol. 2017 Apr 24;8:153. doi: 10.3389/fneur.2017.00153. eCollection 2017. PMID 28484421
- [Result] Ulm L, Ohlraun S, Harms H, Hoffmann S, Klehmet J, Ebmeyer S, Hartmann O, Meisel C, Anker SD, Meisel A. STRoke Adverse outcome is associated WIth NoSocomial Infections (STRAWINSKI): procalcitonin ultrasensitive-guided antibacterial therapy in severe ischaemic stroke patients - rationale and protocol for a randomized controlled trial. Int J Stroke. 2013 Oct;8(7):598-603. doi: 10.1111/j.1747-4949.2012.00858.x. Epub 2012 Aug 28. PMID 22925000
- [Result] Hotter B, Hoffmann S, Ulm L, Montaner J, Bustamante A, Meisel C, Meisel A. Inflammatory and stress markers predicting pneumonia, outcome, and etiology in patients with stroke: Biomarkers for predicting pneumonia, functional outcome, and death after stroke. Neurol Neuroimmunol Neuroinflamm. 2020 Feb 25;7(3):e692. doi: 10.1212/NXI.0000000000000692. Print 2020 May. PMID 32098866
- [Result] Hotter B, Hoffmann S, Ulm L, Meisel C, Bustamante A, Montaner J, Katan M, Smith CJ, Meisel A. External Validation of Five Scores to Predict Stroke-Associated Pneumonia and the Role of Selected Blood Biomarkers. Stroke. 2021 Jan;52(1):325-330. doi: 10.1161/STROKEAHA.120.031884. Epub 2020 Dec 7. PMID 33280547
- [Result] Hotter B, Ulm L, Hoffmann S, Katan M, Montaner J, Bustamante A, Meisel A. Selection bias in clinical stroke trials depending on ability to consent. BMC Neurol. 2017 Dec 4;17(1):206. doi: 10.1186/s12883-017-0989-9. PMID 29202730